CLINICAL TRIAL: NCT05144347
Title: A Dose-Escalation and Expansion Study of the Safety and Pharmacokinetics of XL114 Administered in Subjects With Non-Hodgkin's Lymphoma
Brief Title: Study of XL114 in Subjects With Non-Hodgkin's Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to Sponsor reasons.
Sponsor: Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: XL114-101
Record Dates: First submitted 2021-11-10; First posted 2021-12-03 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Non-Hodgkin's Lymphoma (NHL); Activated B-Cell Type Diffuse Large B-Cell Lymphoma (ABC-DLBCL); Mantle Cell Lymphoma (MCL); Chronic Lymphocytic Leukemia (CLL); Small Lymphocytic Lymphoma (SLL)
Keywords: Mucosa-associated Lymphoid Tissue Lymphoma Translocation Protein 1 (MALT-1); B-cell Malignancies; Fatty Acid Binding Protein 5 (FABP-5)
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Mantle-Cell; Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Intervention Model Description: Dose-escalation followed by Cohort-expansion in NHL-specific expansion cohorts
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- XL114 Dose-Escalation Cohorts (Experimental): Subjects (Cohort A1-An) will accrue in cohorts of 3-12 subjects in a i3+3 design.
  Interventions: Drug: XL114
- XL114 Expansion Cohorts (Experimental): The recommended dose from the Dose-Escalation stage, will be used in subjects with activated B-cell-like diffuse large B-cell lymphoma [ABC-DLBCL] (Cohort B), mantle cell lymphoma [MCL] (Cohort C), chronic lymphocytic leukemia [CLL]/small lymphocytic lymphoma [SLL] (Cohort D). Subjects will also be enrolled in a Biomarker cohort (Cohort E).
  Interventions: Drug: XL114

INTERVENTIONS:
Drug: XL114 — Tablets of XL114

SUMMARY:
This is a Phase 1, non-randomized, open-label, dose-escalation and expansion study, evaluating the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and preliminary clinical antitumor activity of XL114 administered alone orally to subjects with Non-Hodgkin's Lymphoma (NHL). The objectives of the study also include determining the recommended dose (RD) and/or maximum tolerated dose (MTD) of XL114.

ELIGIBILITY:
Inclusion Criteria:

* Dose-Escalation Stage (Cohort A) and Cohort-Expansion Stage (B-E): The subject has received standard life-prolonging therapies or are not qualified to receive such therapies.
* Dose-Escalation Stage (Cohort A): Subjects with histologically documented diagnosis of B-cell or T-cell Non-Hodgkin's Lymphoma as defined by the World Health Organization (WHO) classification. Note: Refer to exclusion criteria for lymphoma subtypes which are excluded from study participation.
* Cohort-Expansion Stage Cohort B (ABC-DLBCL subtype): Subjects with histologically documented activated B-cell diffuse large B-cell lymphoma (ABC-DLBCL) subtype. Note: De novo or transformed diffuse large B-cell lymphoma (DLBCL) from previously diagnosed indolent lymphoma (eg, follicular lymphoma) is allowed.
* Cohort-Expansion Stage Cohort C (MCL): Subjects with histologically documented MCL with monoclonal B-cells that show a chromosome translocation t(11;14)(q13;q32) and/or overexpression of cyclin D1.
* Cohort-Expansion Stage Cohort D (CLL/SLL): Subjects with histologically documented CLL/SLL per the International Workshop on Chronic Lymphocytic Leukemia (iwCLL) guidelines.
* Cohort-Expansion Stage Cohort E, Biomarker Cohort (ABC-DLBCL, MCL, and SLL): Subjects with ABC-DLBCL, MCL, and SLL that fulfill the subject disease characteristics criteria as described for Cohorts B, C, or D.
* Cohort-Expansion Stage: Subjects with ABC-DLBCL, MCL, and SLL must have measurable disease by revised criteria for response assessment of lymphoma.
* Cohort-Expansion Stages: Must have archival tumor tissue available, which was collected up to 2 years prior to consent for this study. If archival tumor tissue is not available, a fresh tumor biopsy may be obtained (if safe to acquire) up to 60 days prior to first dose.
* Biomarker Cohort: Subjects must provide a fresh tumor biopsy up to 60 days prior to first dose, at week 2, day 1 (W2D1) after initiation of XL114, and at disease progression. Note: The tumor tissue requirement in the Expansion and Biomarker cohorts doesn't apply for subjects with CLL.
* Recovery to baseline or ≤ Grade 1 severity (Common Terminology Criteria for Adverse Events version 5 [CTCAE v5]) from AEs, unless AEs are clinically nonsignificant or stable.
* Left ventricular ejection fraction (LVEF) > 50% as determined by echocardiogram (ECHO) or multigated acquisition (MUGA) scan per local standard.
* Age 18 years or older on the day of consent.
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0-1
* Adequate organ and marrow function
* Sexually active fertile subjects and their partners must agree to highly effective methods of contraception.
* Female subjects of childbearing potential must not be pregnant at screening.

Exclusion Criteria:

* Receipt of prior therapies as defined in the protocol
* The following lymphoma types/manifestations are not eligible for this study: Burkitt's lymphoma (BL), Burkitt-like lymphoma (BLL), lymphoblastic lymphoma/leukemia (LBL), post-transplant lymphoproliferative disease (PTLD), primary mediastinal (thymic) large B-cell lymphoma (PMBL), lymphomas involving the central nervous system (CNS) or meninges
* History of autoimmune hemolytic anemia (AIHA) or idiopathic thrombocytopenic purpura (ITP).
* History of solid organ or allogeneic hematopoietic stem cell transplantation.
* Concomitant anticoagulation with the oral anticoagulants apixaban, betrixaban, rivaroxaban, and dabigatran.
* Use of a strong inhibitor or inducer of cytochrome P450 3A4 (CYP3A4) within 5 half-lives or 4 weeks prior to first dose of study treatment, whichever is shorter.
* Uncontrolled, significant intercurrent or recent illness
* Major surgery (eg, GI surgery) within 3 weeks before first dose of study treatment.
* Corrected QT interval calculated by the Fridericia formula (QTcF) > 470 ms per electrocardiogram (ECG).
* Pregnant or lactating females.
* Inability to swallow XL114 tablets.
* Diagnosis of another malignancy within 2 years before first dose of study treatment, except for superficial skin cancers, or localized, low-grade tumors deemed cured and not treated with systemic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-04-12 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Dose-Escalation Stage: Recommended Dose (RD) and/or Maximum Tolerated Dose (MTD) for XL114 | 4-6 months
  To determine the RD and/or MTD of XL114 administered orally in subjects with NHL
Cohort-Expansion Stage: Objective Response Rate (ORR) | 4-6 months
  To evaluate preliminary efficacy of XL114 by estimating the ORR based on lymphoma-specific response criteria as assessed by the Investigator

SECONDARY OUTCOMES:
Safety of XL114, as evaluated by Adverse Events (AEs) | 4-6 months
  To evaluate the safety of XL114 through the evaluation of incidence and severity of treatment emergent nonserious adverse events (AEs) and serious adverse events (SAEs)at each dose level and their relationship to study drug treatment.
Tolerability of XL114, as evaluated by Dose Intensity, Dose Modifications, and Study Discontinuation due to AEs | 4-6 months
  To evaluate the tolerability of XL114 through the evaluation of dose intensity, dose modifications and study treatment discontinuation due to AEs related to XL114.
Dose-Escalation Stage: Time to Maximum Plasma Concentration (Tmax) | 4-6 months
  To evaluate the Tmax of XL114.
Dose-Escalation Stage: Maximum Plasma Concentration (Cmax) | 4-6 months
  To evaluate the Cmax of XL114.
Dose-Escalation Stage: Area Under the Plasma Concentration-Time Curve Over the Last 24-hour Dosing Interval (AUC 0-24) | 4-6 months
  To evaluate the AUC 0-24 of XL114.
Dose-Escalation Stage: Terminal Half-Life | 4-6 months
  To evaluate the terminal half-life of XL114.
Dose-Escalation Stage: Apparent Clearance (CL/F) | 4-6 months
  To evaluate the CL/F of XL114.
Cohort-Expansion Stage: Antitumor Activity of XL114 (Objective Response Rate [ORR]) | 4-6 months
  To evaluate the antitumor activity of XL114 as measured by ORR based on lymphoma-specific response criteria as assessed by a Blinded Independent Radiology Committee (BIRC) for selected cohorts.
Cohort-Expansion Stage: Antitumor Activity of XL114 (Duration of Response [DOR]) | 4-6 months
  To evaluate the antitumor activity of XL114 as measured by DOR based on lymphoma-specific response criteria as assessed by the Investigator or by a Blinded Independent Radiology Committee (BIRC) for selected cohorts.
Cohort-Expansion Stage: Antitumor Activity of XL114 (Progression Free Survival [PFS]) | 4-6 months
  To evaluate the antitumor activity of XL114 as measured by PFS based on lymphoma-specific response criteria as assessed by the Investigator or by a Blinded Independent Radiology Committee (BIRC) for selected cohorts.
Cohort-Expansion Stage: Overall Survival (OS) of XL114 | 4-6 months
  To evaluate duration of overall survival (OS)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Exelixis Clinical Site #3, Tucson, Arizona
  - Exelixis Clinical Site #1, Indianapolis, Indiana
  - Exelixis Clinical #4, Pittsburgh, Pennsylvania
  - Exelixis Clinical Site #2, Spokane, Washington